CLINICAL TRIAL: NCT02127619
Title: Prospective Study of Total Knee Replacement With the ROCC Knee
Brief Title: Total Knee Replacement With the ROCC Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bercovy, Michel, M.D. (Individual)
Responsible Party: Principal Investigator, Dr Bercovy, Orthopedic Surgeon, Bercovy, Michel, M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 602-ROCC
Record Dates: First submitted 2014-04-25; First posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis
Keywords: knee prosthesis; total knee replacement; total knee arthroplasty; prospective study; Therapeutic level IV
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Total knee replacement with the ROCC® knee prosthesis — replacement of an osteoarthritic knee with a total knee prosthesis operation may be for a single knee ( unilateral) or both knees of a patient ( bilateral)
  Other Names: Total knee arthroplasty; Total knee prosthesis

SUMMARY:
The purpose of this study was to assess the results of a Total Knee prosthesis specifically intended to enhance functional performance , especially in terms of physical and sports activity.

DETAILED DESCRIPTION:
Clinical and radiographic results , complications, early post-operative and late functional outcome and survivorship were studied in a continuous prospective series of 500 patients ( 602 knees) managed using the ROCC knee ( BIOMET INC - Warsaw- IND, USA).

A minimum follow-up of 5 years was required.

ELIGIBILITY:
Inclusion Criteria:

* all patients receiving a total knee

Exclusion Criteria:

* patients with severe psychiatric, neurologic, cardiologic or locomotor pathology occuring after the total knee replacement

Ages: 42 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2001-01; Primary Completion 2008-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
locomotor function with the Knee society score | at a minimum of 5 years after surgery

SECONDARY OUTCOMES:
physical and sports activities with the UCLA activity score | at last follow-up examination, with minimum of 5 years after surgery
clinical status with the Oxford Knee Score | before surgery
clinical status with the Oxford knee score | at last follow-up examination, with minimum of 5 years after surgery
WOMAC ARTHRITIS INDEX | before surgery
WOMAC ARTHRITIS INDEX | at last follow-up examination, with minimum of 5 years after surgery

OTHER OUTCOMES:
patient satisfaction with the Forgotten Joint Score | at last follow-up examination, with minimum of 5 years after surgery
  this score asseses the perfection on patient's point of view for a total knee replacement
positioning and quality of the fixation of a total knee replacement | minimum 5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bercovy, md, Principal Investigator — Clinique Les Fontaines- 77000 - Melun- FRANCE
Locations (1):
- Clinique Les Fontaines, Melun, France